CLINICAL TRIAL: NCT02228408
Title: A Phase IV Randomized, Double-blind, Active-controlled, Single-center Study of the Safety and Effects on Cardiac Structure and Function of Hydralazine and Isosorbide Dinitrate in Patients With Hemodialysis Dependent ESRD
Brief Title: Safety and Cardiovascular Efficacy of Hydralazine and Isosorbide Dinitrate in Dialysis-Dependent ESRD
Acronym: HIDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Charytan M.D., Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DK100772-01
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Chronic Hemodialysis (ESRD)
Keywords: hemodialysis; ESRD; Cardiovascular Disease; Isosorbide Dinitrate; Hydralazine
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases | interventions — Hydralazine; Isosorbide Dinitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydralazine/Isorsorbide Dinitrate (Experimental): Hydralazine/Isorsorbide Dinitrate (ISD/HY) will be administered with a target dose of 40 mg of ISD and 75 mg of Hydralazine 3x/daily. Doses will be titrated between weeks 0-4 and may be decreased as necessary for treatment of adverse events.
  Allowable Dosage Forms:
  ISD/HY 10 mg/10-3x/day ISD/HY 20 mg/35mg-3x/day ISD/HY 40 mg/75 mg-3x/day
  Interventions: Drug: Hydralazine/Isorsorbide Dinitrate
- Placebo (Active Comparator): Placebo will be administered Doses will be titrated between weeks 0-4 and may be decreased as necessary for treatment of adverse events.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydralazine/Isorsorbide Dinitrate — Hydralazine/Isorsorbide Dinitrate (ISD/HY) will be administered with a target dose of 40 mg of ISD and 75 mg of Hydralazine 3x/daily. Doses will be titrated between weeks 0-4 and may be decreased as necessary for treatment of adverse events.
  Target Dose:
  Hydralazine 75 mg 3x day Isorsorbide Dintrate 40 mg 3x/day
  Allowable Dosage Forms:
  ISD/HY 10 mg/10-3x/day ISD/HY 20 mg/35 mg-3x/day ISD/HY 40 mg/75 mg-3x/day
  Dose Titration:
  ISD/HY will be administered at a starting dose ISD/HY 10 mg/10-3x/day and titrated to ISD/HY 20 mg/35 mg-3x/day after 4 days and to ISD/HY 40 mg/75 mg-3x/day at 4 weeks. Dose will be decreased as necessary for dose-limiting side effects.
  Other Names: Apresoline; Isordil
  Arms: Hydralazine/Isorsorbide Dinitrate
Drug: Placebo — Placebo titration will mimic titration of active study arm
  Arms: Placebo

SUMMARY:
This study is a pilot study designed to compare the safety and cardiovascular effects of 26 weeks of combination hydralazine/isorsorbide dinitrate therapy with placebo therapy in patients receiving chronic hemodialysis.

The investigators hypothesize that treatment of chronic hemodialysis (ESRD) patients with a combination of hydralazine/isosorbide dinitrate compared with placebo is safe and that it will improve heart function as well blood flow/blood vessel supply.

DETAILED DESCRIPTION:
Sixteen patients receiving maintenance hemodialysis will be randomized to 26 weeks of therapy with combination hydralazine/isosorbide dinitrate or placebo. Study medications will be titrated to goal dose during the first 4 weeks and maintained at goal dose (as tolerated) between weeks 4-26. A final study visit to assess symptoms after drug discontinuation will occur 4 weeks after drug discontinuation.

Study duration-Maximum of 32 weeks with 26 weeks of active therapy.

Efficacy Measures -Tissue Doppler echocardiography and myocardial perfusion scanning using radioactive NH3 PET will be assessed at weeks 0 and 26.

Safety Measures-Adverse events rates including inter- and intra-dialytic hypotension, ,cardiovascular death and gastrointestinal symptoms will be assessed throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria

1. Maintenance hemodialysis therapy for end-stage renal disease
2. Age 18-85 years
3. ≥ 90 days since dialysis initiation
4. Ability to provide informed consent
5. Pre-dialysis seated systolic blood pressure measurements must be ≥ 120 mm Hg in the 2 weeks before enrollment and on the day of randomization.

Exclusion Criteria

1. Serum potassium ≥6.5 mEq/L within 2 months prior to screening
2. Unscheduled dialysis for hyperkalemia within the 3 months prior to screening
3. Hypotension defined as pre-dialysis SBP <100 mm Hg (seated measurement) within 4 weeks prior to enrollment
4. Recurrent intra-dialytic hypotension, defined as systolic blood pressure <80 mm Hg during ≥3 dialysis sessions per 30-day rolling period or treatment for either hypotension or symptoms of hypotension if systolic blood pressure is < 100 mm Hg during ≥3 dialysis sessions per 30-day rolling period.
5. Mitral valve repair or replacement
6. Severe mitral valve disease by echocardiography, coronary angiography or cardiac magnetic resonance imaging
7. Prior coronary artery bypass graft
8. Anticipated kidney transplant, change to peritoneal dialysis, or transfer to another dialysis unit within 6 months
9. Expected survival < 6 months
10. Allergy to study medications (ISD, HY, adenosine/diprimidole)
11. Active use of sildenafil, vardenafil or tadalafil
12. History of severe aortic stenosis or other cause of LV outflow obstruction
13. Pregnancy, anticipated pregnancy, or breastfeeding, confirmed by serum pregnancy test on the day of PET scan
14. Incarceration
15. Participation in another intervention study
16. Use of monoamine oxidase inhibitors
17. Contraindication to adenosine including

    * 2nd or 3rd degree heart block, sick sinus syndrome or symptomatic bradycardia (without a functioning pacemaker)
    * moderate or severe asthma
    * chronic obstructive pulmonary disease
18. Active use of any of the study medications unless participant and physician willing to discontinue prior to enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Charytan, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
deidentified may be shared upon request to the PI

REFERENCES:
- [Derived] Mugendi GA, Mutua FM, Natale P, Esterhuizen TM, Strippoli GF. Calcium channel blockers for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 Oct 1;10(10):CD011064. doi: 10.1002/14651858.CD011064.pub2. PMID 33000470

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydralazine/Isorsorbide Dinitrate: Hydralazine/Isorsorbide Dinitrate (ISD/HY) will be administered with a target dose of 40 mg of ISD and 75 mg of Hydralazine 3x/daily. Doses will be titrated between weeks 0-4 and may be decreased as necessary for treatment of adverse events.
  Allowable Dosage Forms:
  ISD/HY 10 mg/10-3x/day ISD/HY 20 mg/35mg-3x/day ISD/HY 40 mg/75 mg-3x/day
  Hydralazine/Isorsorbide Dinitrate: Hydralazine/Isorsorbide Dinitrate (ISD/HY) will be administered with a target dose of 40 mg of ISD and 75 mg of Hydralazine 3x/daily. Doses will be titrated between weeks 0-4 and may be decreased as necessary for treatment of adverse events.
  Target Dose:
  Hydralazine 75 mg 3x day Isorsorbide Dintrate 40 mg 3x/day
  Allowable Dosage Forms:
  ISD/HY 10 mg/10-3x/day ISD/HY 20 mg/35 mg-3x/day ISD/HY 40 mg/75 mg-3x/day
  Dose Titration:
  ISD/HY will be administered at a starting dose ISD/HY 10 mg/10-3x/day and titrated to ISD/HY 20 mg/35 mg-3x/day after 4 days and to ISD/HY 40 mg/75 mg-3x/day at 4 weeks. Dose will be decreased as necessary for dose-limiting side effects.
Period: Overall Study
Arm/Group | Hydralazine/Isorsorbide Dinitrate | Placebo
Started | 7 | 10
Completed | 7 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydralazine/Isorsorbide Dinitrate | Placebo | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [54 to 65] | 63 [55 to 68] | 62 [53 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Rate of Hypotension, Serious Adverse Events, GI Events and Cardiovascular Death
Description: Rate of primary Safety Outcomes(hypotension, serious adverse events, GI events and CV death)
Time Frame: 6 months
Population: intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Hydralazine/Isorsorbide Dinitrate | Placebo
Number analyzed (Participants) | 7 | 10
Participants
  intradialytic hpypotension | 1 | 6
  SAE | 5 | 3
  Nausea | 4 | 3
  CV death rate per patient year | 0 | 0
Statistical Analysis 1: Comparison: Hydralazine/Isorsorbide Dinitrate vs Placebo; Test type: Superiority; p = 0.04, poisson

2. Primary Outcome: Efficacy-Change in Coronary Flow Reserve (CFR) From 0-6 Months
Description: Primary Efficacy Measure-CFR measured on rest and stress Positron Emission Tomography
Time Frame: 0 to 6 months
Population: intent to treat
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Hydralazine/Isorsorbide Dinitrate | Placebo
Number analyzed (Participants) | 6 | 10
ratio | -0.27 (0.23) | -0.03 (0.46)
Statistical Analysis 1: Comparison: Hydralazine/Isorsorbide Dinitrate vs Placebo; Test type: Superiority; p = 0.19, t-test, 2 sided

3. Primary Outcome: Change in E' on TDI Echo From 0-6 Months
Description: Co-primary efficacy measure measured on Tissue Doppler Echocardiography
Time Frame: 0 to 6 months
Population: intent to treat
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Hydralazine/Isorsorbide Dinitrate | Placebo
Number analyzed (Participants) | 6 | 10
cm/s | 0.56 (1.1) | -0.04 (0.92)
Statistical Analysis 1: Comparison: Hydralazine/Isorsorbide Dinitrate vs Placebo; Test type: Superiority; p = 0.34, t-test, 2 sided

4. Primary Outcome: Reduction in Drug Dose or Discontinuation of Study Drug
Description: Primary Tolerability measure
Time Frame: 0 to 6 months
Population: intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Hydralazine/Isorsorbide Dinitrate | Placebo
Number analyzed (Participants) | 7 | 10
Participants
  discontinuation | 0 | 0
  reduction | 2 | 3

5. Primary Outcome: Number of Patients Completing Study From 0 to 6 Months
Description: Primary Feasibility Measure
Time Frame: 0 to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hydralazine/Isorsorbide Dinitrate | Placebo
Number analyzed (Participants) | 7 | 10
Participants | 6 | 10

6. Secondary Outcome: Change in Circulating Fibrosis Markers and Angiogenesis Markers
Description: Circulating concentrations of markers such as the carboxy terminal of pro-collagen type 1 or ADMA will be measured
Time Frame: 0 to 6 months
Population: Not done-data. samples not analyzed due to lack of additional funding.
Arm/Group | Hydralazine/Isorsorbide Dinitrate | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in LVMI
Description: Change in left ventricular mass index between baseline and 6 months.
Time Frame: 0 to 6 months
Measure: Mean (Standard Deviation); unit: g/m2
Arm/Group | Hydralazine/Isorsorbide Dinitrate | Placebo
Number analyzed (Participants) | 6 | 10
g/m2 | -10.6 (8.5) | -8 (11.1)
Statistical Analysis 1: Comparison: Hydralazine/Isorsorbide Dinitrate vs Placebo; Test type: Superiority; p = 0.62, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Hydralazine/Isorsorbide Dinitrate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 5/7 | 3/10
Other Adverse Events (participants affected / at risk) | 7/7 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydralazine/Isorsorbide Dinitrate (N=7) | Placebo (N=10)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
cv hospitalization (Cardiac disorders) | 1 (1) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
av fisula thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
gi bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydralazine/Isorsorbide Dinitrate (N=7) | Placebo (N=10)
diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
headache (Gastrointestinal disorders) | 5 (8) | 7 (7)
vomitting (Gastrointestinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
small study. unbalanced randomization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT02228408/Prot_SAP_000.pdf